CLINICAL TRIAL: NCT03449160
Title: Addition of Postural Training Device (UPRIGHT) to Routine Physical Therapy for the Treatment of Back Pain: a Randomized Trial
Brief Title: Postural Training Device (UPRIGHT) for Back Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID 19 which is preventing outpatient and elective procedures
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Byron Schneider, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSCHNEIDERXX
Record Dates: First submitted 2018-01-04; First posted 2018-02-28 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Back Pain Without Radiation; Back Pain, Low
MeSH Terms: conditions — Back Pain; Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Therapy (Active Comparator): Receive standard physical therapy
  Interventions: Other: physical therapy
- posture training device (Experimental): Receive a posture training device in addition to standard physical therapy
  Interventions: Device: UPRIGHT

INTERVENTIONS:
Device: UPRIGHT — A small externally wearable device that is placed on the back, which gently vibrates when correct posture is not maintained. The device is removable, and used for only portions of the day
  Arms: posture training device
Other: physical therapy — routine physical therapy
  Arms: Physical Therapy

SUMMARY:
Participants with low back pain who are referred for physical therapy will be randomized to routine physical therapy or routine physical therapy plus receiving a postural training device

DETAILED DESCRIPTION:
Participants with low back pain who are referred for physical therapy will be randomized to routine physical therapy or routine physical therapy plus receiving a postural training device.

Physical therapy will be completed 1-2 times per week over 4-6 weeks. If randomized to the group that also receives a postural training device, one of the physical therapy sessions will instruct the patient on use of the device, which can be used thereafter as tolerated by the patient.

At 6 weeks and 3 months, questionnaires that assess patients pain and function will be completed to assess outcomes

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65, capable of understanding and providing consent in English, capable of complying with the outcome instruments used, and capable of attending all planned therapy sessions
* Primary complaint of lumbar or thoracic pain thought to be at least in part due to mechanical/postural etiologies based on clinical presentation
* 7 day average numeric pain rating score (NPRS) of at least 4 on a 0-10 scale at baseline evaluation
* Pain duration of at least 2 months
* Patient owns and is familiar with the use of a personal smart phone
* Patient consents to treatment with postural based physical therapy. In order to maintain blinding, patients will not be provided with details of the treatment plan until after the randomization process has been performed. They will only be informed of the treatment protocol for the group to which they have been assigned.

Exclusion Criteria:

* *History of prior thoracic or lumbar fusion surgery

  * Acute Spine fracture
  * Current pregnancy
  * BMI over 40
  * Inability to sense UPRIGHT vibration
  * Active Systemic inflammatory arthritis (e.g. rheumatoid arthritis, ankylosing spondylitis, lupus)
  * Medical conditions causing significant functional disability (e.g. stroke, spinal cord injury, amputation)
  * Severe Chronic widespread pain or somatoform disorder (e.g. fibromyalgia)
  * Severe clinical depression, or psychotic features
  * Implanted electrical medical device (i.e. cardiac pacemaker/defibrillator, spinal cord stimulator, bladder stimulator)
  * Allergic skin reaction to tapes or adhesives
  * Worker's compensation claim or legal action related to the thoracic or lumbar pain
  * Patients unable to read English and complete the assessment instruments
  * Patients unable to attend assigned physical therapy sessions
  * Incarcerated patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Improvement/Change in Pain | Primary outcome is at 6 weeks, secondary time point 12 weeks
  0-10 pain scale

SECONDARY OUTCOMES:
Improvement/Change Disability | 6 weeks, 12 weeks
  Modified Oswestry Disability Index

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No